CLINICAL TRIAL: NCT03164993
Title: ALICE: a Randomized Placebo-controlled Phase II Study Evaluating Atezolizumab Combined with Immunogenic Chemotherapy in Patients with Metastatic Triple-negative Breast Cancer
Brief Title: Atezolizumab Combined with Immunogenic Chemotherapy in Patients with Metastatic Triple-negative Breast Cancer
Acronym: ALICE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Collaborators: Hoffmann-La Roche (Industry); Norwegian Cancer Society (Other); St. Olavs Hospital (Other); Helse Stavanger HF (Other Government); Rigshospitalet, Denmark (Other); Vejle Hospital (Other); NanoString Technologies, Inc. (Industry); Technical University of Denmark (Other); Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Jon Amund Kyte, National coordinating investigator, Oslo University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ML39079_ALICE
Record Dates: First submitted 2017-05-12; First posted 2017-05-24 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2023-10

CONDITIONS: Cancer, Breast; Triple Negative Breast Cancer
Keywords: Neoplasms
MeSH Terms: conditions — Breast Neoplasms; Triple Negative Breast Neoplasms; Neoplasms | interventions — atezolizumab; liposomal doxorubicin; Cyclophosphamide

STUDY DESIGN:
Intervention Model Description: Randomized, double-blind, placebo-controlled
Who Masked: Participant, Investigator
Masking Description: Randomization will be performed using the eCRF. The subject will allocated to a randomization number and the randomization number will be sent to the hospital pharmacy. The pharmacy keeps the randomization listing and prepares the infusion according to the given randomization number. The pharmacy will keep a log of all infusions prepared. All other study personell will be blinded to the treatment code.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm Chemotherapy + Placebo (Placebo Comparator): Chemo (pegylated liposomal doxorubicin + cyclophosphamide) + placebo
  Interventions: Drug: Pegylated liposomal doxorubicin; Drug: Cyclophosphamide; Other: Placebo
- Arm Chemotherapy + Atezolizumab (Active Comparator): Chemo (pegylated liposomal doxorubicin + cyclophosphamide) + Atezolizumab
  Interventions: Drug: Atezolizumab; Drug: Pegylated liposomal doxorubicin; Drug: Cyclophosphamide

INTERVENTIONS:
Drug: Atezolizumab — Atezolizumab is a monoclonal antibody designed to target and bind to a protein called PD-L1 (programmed death ligand-1), which is expressed on tumour cells and tumour-infiltrating immune cells. PD-L1 interacts with PD-1 and B7.1, both found on the surface of T cells, causing inhibition of T cells. By blocking this interaction, Atezolizumab may enable the activation of T cells, restoring their ability to effectively detect and attack tumour cells.
  Other Names: Tecentriq
  Arms: Arm Chemotherapy + Atezolizumab
Drug: Pegylated liposomal doxorubicin — Chemotherapy
Drug: Cyclophosphamide — Chemotherapy
Other: Placebo — Placebo
  Arms: Arm Chemotherapy + Placebo

SUMMARY:
This is a randomized, double-blind, placebo-controlled phase II study evaluating the safety and efficacy of Atezolizumab when combined with immunogenic chemotherapy in subjects with metastatic triple-negative breast cancer. Atezolizumab, pegylated liposomal doxorubicin and cyclophosphamide are the Investigational Medicinal Products (IMPs).

DETAILED DESCRIPTION:
Breast cancer is rarely curable after metastasis, and the therapeutic options for metastatic triple negative breast cancer (TNBC) are limited. The host immune response is strongly predictive for the effect of chemotherapy in patients with TNBC. In the present trial, we combine Atezolizumab, an inhibitory antibody against Programmed Death Ligand-1 (PD-L1), with chemotherapy. Thereby, we aim to release the brake on the chemo-induced immune response. The chemotherapeutic regime is a combination of anthracycline and cyclophosphamide, applied in a semi-metronomic fashion (pegylated liposomal doxorubicin every 2nd week and daily cyclophosphamide for 2/4 weeks). The investigators hypothesize that the semi-metronomic regime will induce immunological cell death and counter T regulatory cells, while maintaining the leukocyte counts and the ability of the effector immune cells to respond. The use of pegylated liposomal doxorubicin (Caelyx) minimizes the adverse effects of anthracyclines on the heart and allows for continued treatment beyond the otherwise mandatory anthracycline limits.

ELIGIBILITY:
Inclusion Criteria:

1. Metastatic or incurable locally advanced, histologically documented TNBC (negative for HER2, ER and PR ). HER2 negativity is defined as either of the following by local laboratory assessment: In situ hybridization (ISH) non-amplified (ratio of HER2 to CEP17 < 2.0 or single probe average HER2 gene copy number < 4 signals/cell), or IHC 0 or IHC 1+ (if more than one test result is available and not all results meet the inclusion criterion definition, all results should be discussed with the PI to establish eligibility of the patient). ER and PR negativity are defined as < 1% and <10%, respectively, of cells expressing hormonal receptors via IHC analysis
2. Adequate newly obtained core or excisional biopsy of a tumor lesion not previously irradiated. No anti-tumor treatment is allowed between the time point for biopsy and study entry. If a patient has undergone chemotherapy in the metastatic setting, a new biopsy must be obtained after this therapy
3. Measurable disease according to iRECIST
4. Signed Informed Consent Form
5. Women or men aged ≥ 18 years
6. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
7. In patients that have received (neo)adjuvant treatment with anthracyclines or cyclophosphamide, a minimum of 12 months from treatment with anthracyclines or cyclophosphamide until relapse of disease is required
8. A maximum of one previous line with chemotherapy in the metastatic setting
9. Female subject of childbearing potential should have a negative urine or serum pregnancy test within 7 days prior to receiving the first dose of study medication. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required
10. Female subjects of childbearing potential should agree to remain abstinent (refrain from heterosexual intercourse) or use contraceptive methods that result in a failure rate of < 1% per year, during the treatment period and for at least 5 months after the last dose of study therapy. A woman is considered to be of childbearing potential if she is postmenarcheal, has not reached a postmenopausal state (≥ 12 continuous months of amenorrhea with no identified cause other than menopause), and has not undergone surgical sterilization (removal of ovaries and/or uterus). Examples of contraceptive methods with a failure rate of < 1% per year include bilateral tubal ligation, male sterilization, proper use of hormonal contraceptives that inhibit ovulation and hormone-releasing intrauterine devices (IUDs). Periodic abstinence (e.g., calendar, ovulation, symptothermal, or postovulation methods) and withdrawal are not acceptable methods of contraception
11. Male subjects should agree to use an adequate method of contraception starting with the first dose of study therapy through 3 months after the last dose of study therapy
12. Able to swallow orally administrated medication.
13. Adequate organ function as defined in Table 1 in the protocol.

Exclusion Criteria:

1. Malignancies other than breast cancer within 5 years prior to randomization, with the exception of those with a negligible risk of metastasis or death and treated with expected curative outcome (such as adequately treated carcinoma in situ of the cervix or basal or squamous cell skin cancer)
2. Patients with known PD-L1 positive TNBC, as assessed by the Ventana SP142 assay (IC ≥1%), and no previous chemotherapy in the metastatic setting, should be offered standard therapy with nab-paclitaxel/atezolizumab outside of the trial, if they had a disease free interval of >12 months after previous (neo)adjuvant chemotherapy, unless the patient for other reasons should not receive nab-paclitaxel, according to own preferences, drug availability or recommendations by the treating physician. A history of progression on taxanes in the neoadjuvant setting, or severe side effects from taxane therapy, may represent sufficient reason to offer the patient inclusion into the the ALICE-trial, if the physician considers that the patient should receive antracyclines rather than taxanes as 1st line therapy for metastatic disease. If more than one TNBC biopsy has been evaluated for PD-L1 by the SP142 assay, and the results differ, the patient's PD-L1 status determination will be based on best clinical judgment.
3. Spinal cord compression not definitively treated with surgery and/or radiation, or previously diagnosed and treated spinal cord compression without evidence that disease has been clinically stable for > 2 weeks prior to randomization
4. Known CNS disease, except for asymptomatic CNS metastases, provided all of the following criteria are met:

   1. Measurable disease outside the CNS
   2. No metastases to mesencephalon, pons, medulla oblongata, or spinal cord
   3. No ongoing requirement for dexamethasone as therapy for CNS disease
   4. No radiation of brain lesions within 7 days prior to randomization
   5. No leptomeningeal disease
   6. Patients with symptomatic CNS metastases must receive radiation therapy and/or surgery for CNS metastases. Following treatment, these patients may be eligible, if all other criteria are met
5. Uncontrolled pleural effusion, pericardial effusion, or ascites. Patients with indwelling catheters (e.g., PleurX®) are allowed
6. Uncontrolled tumor-related pain. Patients requiring narcotic pain medication must be on a stable regimen at study entry. Symptomatic lesions (e.g., bone metastases or metastases causing nerve impingement) amenable to palliative radiotherapy should be treated prior to randomization. Asymptomatic metastatic lesions whose further growth would likely cause functional deficits or intractable pain (e.g., epidural metastasis that is not presently associated with spinal cord compression) should be considered for loco-regional therapy if appropriate prior to randomization
7. Ionized calcium > 1.2 x UNL. The use of bisphosphonates is allowed
8. Pregnant or breastfeeding
9. Evidence of significant uncontrolled concomitant disease that could affect compliance with the protocol or interpretation of results, including significant liver disease (such as cirrhosis, uncontrolled major seizure disorder, or superior vena cava syndrome)
10. Significant cardiovascular disease, such as New York Heart Association (NYHA) cardiac disease (Class II or greater), myocardial infarction within 3 months prior to randomization, unstable arrhythmias, or unstable angina. Patients with a known left ventricular ejection fraction (LVEF) < 40% will be excluded. Patients with known coronary artery disease, congestive heart failure not meeting the above criteria, or LVEF < 50% must be on a stable medical regimen that is optimized in the opinion of the treating physician, in consultation with a cardiologist if appropriate
11. Severe infection within 14 days prior to randomization, requiring hospitalization
12. Received oral or IV antibiotics within 1 week prior to Cycle 1, Day 1. Patients receiving routine antibiotic prophylaxis (e.g., to prevent chronic obstructive pulmonary disease exacerbation or for dental extraction) are eligible
13. Major surgical procedure within 14 days prior to randomization or anticipation of the need for a major surgical procedure during the course of the study other than for diagnosis. Placement of central venous access catheter(s) is not considered a major surgical procedure and is therefore permitted
14. A history of severe allergic, anaphylactic, or other hypersensitivity reactions to chimeric or humanized antibodies or fusion proteins
15. Known hypersensitivity or allergy to biopharmaceuticals produced in Chinese hamster ovary cells or any component of the atezolizumab formulation
16. Known hypersensitivity to doxorubicin or cyclophosphamide or any of their excipients
17. A history of autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (e.g., thyroxin, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment. Patients with eczema, psoriasis, lichen simplex chronicus or vitiligo with dermatologic manifestations only (e.g., no psoriatic arthritis) are permitted provided that they meet all of the following conditions:

    1. Rash must cover less than 10% of body surface area.
    2. Disease is well controlled at baseline and only requiring low potency topical steroids
    3. No acute exacerbations of underlying condition within the last 12 months (not requiring PUVA [psoralen plus ultraviolet A radiation], methotrexate, retinoids, biologic agents, oral calcineurin inhibitors, high potency or oral steroids)
18. Undergone allogeneic stem cell or solid organ transplantation
19. A history of idiopathic pulmonary fibrosis (including pneumonitis) drug-induced pneumonitis, organizing pneumonia (i.e., bronchiolitis obliterans, cryptogenic organizing pneumonia), or evidence of active pneumonitis on screening chest CT scan. History of radiation pneumonitis in the radiation field (fibrosis) is permitted
20. A positive test for HIV
21. Active hepatitis B (defined as having a positive hepatitis B surface antigen [HBsAg] test at screening) or hepatitis C. Patients with past hepatitis B virus (HBV) infection or resolved HBV infection (defined as having a negative HBsAg test and a positive antibody to hepatitis B core antigen [anti-HBc] antibody test) are eligible. Patients positive for hepatitis C virus (HCV) antibody are eligible only if polymerase chain reaction (PCR) is negative for HCV RNA
22. Active tuberculosis
23. Currently receiving study therapy or has participated in a study of an investigational agent and received study therapy or used an investigational device within 4 weeks of the first dose of treatment
24. Received treatment with immune checkpoint modulators, including anti-CTLA-4, anti-PD-1, or anti-PD-L1 therapeutic antibodies
25. Received treatment with systemic immunostimulatory agents (including but not limited to interferons or IL-2) within 4 weeks or five half-lives of the drug (whichever is shorter) prior to randomization
26. Received treatment with systemic corticosteroids or other systemic immunosuppressive medications (including but not limited to prednisone, dexamethasone, cyclophosphamide, azathioprine, methotrexate, thalidomide, and anti-tumor necrosis factor [TNF] agents) within 2 weeks prior to randomization, or anticipated requirement for systemic immunosuppressive medications during the trial

    1. Patients who have received acute, low-dose, systemic immunosuppressant medications (e.g., a one-time dose of dexamethasone for nausea) may be enrolled in the study
    2. Patients with a history of allergic reaction to IV contrast requiring steroid pre-treatment should have baseline and subsequent tumor assessments performed using MRI
    3. The use of inhaled corticosteroids for chronic obstructive pulmonary disease, mineralocorticoids (e.g., fludrocortisone) for patients with orthostatic hypotension, and low-dose supplemental corticosteroids for adrenocortical insufficiency are allowed
27. Received anti-cancer therapy (medical agents or radiation) within 1 week prior to study Cycle 1, Day 1.
28. A history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating Investigator
29. Known psychiatric or substance abuse disorders that would interfere with cooperation and the requirements of the trial
30. Any reason why, in the opinion of the investigator, the patient should not participate. This includes a careful evulation of whether standard therapy is preferable to the study therapy, for the individual patient.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2023-04-25 (Actual); Study Completion 2023-09-30 (Actual)

PRIMARY OUTCOMES:
Assessment of toxicity of combined treatment with Atezolizumab, pegylated liposomal doxorubicin and cyclophosphamide | From inclusion until last follow-up visit (12 weeks after end of treatment if progressive disease; 12 months after end of treatment if no disease progression)
  Incidence, nature, and severity of adverse events graded according to NCI CTCAE v4.0 and Adverse Event of Special Interest (AESIs) for Atezolizumab
Progression-free survival (PFS) | 3 years
  Descriptive comparison of the PFS rates in the total per protocol (PP) population, and the PD-L1+ PP population

SECONDARY OUTCOMES:
Objective tumor response rate | 3 years
  Assessment of clinical response
Overall survival | 5 years
  Assessment of clinical response
Duration of response | 3 years
  Assessment of clinical response
Durable tumor response rate (DRR; >6 months) | 3 years
  Assessment of clinical response
Patient reported outcome Farigue | 3 years
  Measured by the Chalder Fatigue Questionnaire (FQ)
Patient reported outcome NRS | 3 years
  11 point Numerical Rating Scale (NRS) for pain intensity
Patient reported outcome QLQ-C15-PAL | 3 years
  EORTC quality of life questionnaire (QLQ-C15-PAL)
Assessment of changes in the immunological milieu in tumor and peripheral blood | 3 years
  Considering each study arm separately, and by comparing arm A to arm B
Clinical benefit rate | 3 years
  Assessment of clinical response
Assessment of PD-L1 expression, mutation load and immune gene expression | 3 years
  Biomarkers for clinical response

OTHER OUTCOMES:
Assessment of immunological response | 3 years
  immunological response
Identification of novel and integrated biomarkers | 3 years
  For clinical response, toxicity and immune response
Characterization of tumor evolution induced by the study therapy | 3 years
  Considering each study arm separately, and by comparing arm A to arm B
Characterization of changes in microbiota induced by the study therapy | 3 years
  considering each study arm separately, and by comparing arm A to arm B

CONTACTS AND LOCATIONS:
Overall Officials: Jon Amund Kyte, M.D.-Ph.D., Principal Investigator — Oslo University Hospital
Locations (5):
- Denmark (2):
  - Rigshospitalet, Copenhagen
  - Vejle Sygehus, Vejle
- Norway (3):
  - Oslo University Hospital, Oslo
  - Stavanger University Hospital, Stavanger
  - St. Olavs Hospital, Trondheim

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rossevold AH, Andresen NK, Bjerre CA, Gilje B, Jakobsen EH, Raj SX, Falk RS, Russnes HG, Jahr T, Mathiesen RR, Lomo J, Garred O, Chauhan SK, Lereim RR, Dunn C, Naume B, Kyte JA. Atezolizumab plus anthracycline-based chemotherapy in metastatic triple-negative breast cancer: the randomized, double-blind phase 2b ALICE trial. Nat Med. 2022 Dec;28(12):2573-2583. doi: 10.1038/s41591-022-02126-1. Epub 2022 Dec 8. PMID 36482103
- [Derived] Svalheim KG, Andresen NK, Bjerre C, Gilje B, Jakobsen EH, Falk RS, Naume B, Kaasa S, Kyte JA. Patient-reported outcomes from the randomized ALICE trial evaluating the addition of atezolizumab to anthracycline-based chemotherapy in metastatic triple-negative breast cancer. Breast. 2026 Jan 19;86:104704. doi: 10.1016/j.breast.2026.104704. Online ahead of print. PMID 41581361
- [Derived] Kyte JA, Rossevold A, Falk RS, Naume B. ALICE: a randomized placebo-controlled phase II study evaluating atezolizumab combined with immunogenic chemotherapy in patients with metastatic triple-negative breast cancer. J Transl Med. 2020 Jun 23;18(1):252. doi: 10.1186/s12967-020-02424-7. PMID 32576225